CLINICAL TRIAL: NCT00695929
Title: Levosimendan in Congenital Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: MONA MOMENI, Cliniques Universitaires saint Luc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Levosimendan
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Congenital Cardiovascular Defects; Low Cardiac Output Syndrome
Keywords: cardiac surgery with cardiopulmonary bypass
MeSH Terms: conditions — Cardiac Output, Low | interventions — Simendan; Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Levosimendan — Intravenous injection
Drug: Milrinone — Intravenous injection

SUMMARY:
Many pediatric patients undergoing cardiac surgery under cardiopulmonary bypass for repair of complex congenital malformations, require inotropic support for low cardiac output syndrome. Milrinone through its positive inotropic and vasodilatory effects is widely used for this purpose. The aim of the study is to compare Milrinone with Levosimendan, a novel inotope with calcium-sensitizing properties. We hypothesized that using Levosimendan would result in reduced serum lactate through a higher cardiac index.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing complex cardiac surgery under cardiopulmonary bypass and requiring inotropic support

Exclusion Criteria:

* Patients with renal and/or hepatic dysfunction
* Patients requiring inotropic support before their surgery
* Septic patients

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
serum lactate | 12 h postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium

REFERENCES:
- [Background] De Hert SG, Lorsomradee S, Cromheecke S, Van der Linden PJ. The effects of levosimendan in cardiac surgery patients with poor left ventricular function. Anesth Analg. 2007 Apr;104(4):766-73. doi: 10.1213/01.ane.0000256863.92050.d3. PMID 17377079
- [Background] Namachivayam P, Crossland DS, Butt WW, Shekerdemian LS. Early experience with Levosimendan in children with ventricular dysfunction. Pediatr Crit Care Med. 2006 Sep;7(5):445-8. doi: 10.1097/01.PCC.0000235251.14491.75. PMID 16885788
- [Result] Turanlahti M, Boldt T, Palkama T, Antila S, Lehtonen L, Pesonen E. Pharmacokinetics of levosimendan in pediatric patients evaluated for cardiac surgery. Pediatr Crit Care Med. 2004 Sep;5(5):457-62. doi: 10.1097/01.pcc.0000137355.01277.9c. PMID 15329162